CLINICAL TRIAL: NCT01782404
Title: Open Prospective Study on Reduction of Bacteriuria Following Bladder Irrigation With Chlorhexidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC-0008
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Bacteriuria, Intermittent Catheterization
MeSH Terms: conditions — Bacteriuria

ARMS (1):
- Chlorhexidine (Experimental)
  Interventions: Device: Chlorhexidine

INTERVENTIONS:
Device: Chlorhexidine — Bladder irrigation with chlorhexidine 0.2 mg/ml twice daily

SUMMARY:
This a prospective, non-controlled, open, multi-center study evaluating the reduction of bacteriuria after bladder irrigation with chlorhexidine in spinal cord injured patients with chronic bacteriuria practicing intermittent catheterisation (IC). Patients will be treated with chlorhexidine for bladder irrigation twice daily for a maximum of 7 days.

The study hypothesis is that bladder irrigation with chlorhexidine is efficient for a short term reduction of bacteriuria in patients performing intermittent catheterization (IC).

ELIGIBILITY:
Inclusion Criteria

1. Provision of informed consent
2. Female or male spinal cord injured subject aged 18 years and over
3. Bacteriuria of >10^5 CFU/mL of >1 bacterial species verified during screening visit
4. Regular users of intermittent catheterisation as primary method for bladder management (defined as a normal catheterisation frequency of at least 3 times daily for at least 1 month)
5. Ability to retain fluid in the bladder (approx. 120 ml) for at least 10 minutes, as judged by the investigator

Exclusion Criteria

1. Signs or symptoms of symptomatic UTI that requires treatment, as judged by the investigator.
2. Ongoing antibiotic treatment
3. Known anatomical pathology of the urinary tract that could compromise results, as judged by investigator
4. Subject with severe catheterisation difficulties, as judged by investigator
5. Known hypersensitivity to chlorhexidine
6. Use of other instillation products
7. Pregnancy
8. Use of medications that may affect the bacterial culture in the urine and bladder (e.g. methenamine hippurate)
9. Involvement in the planning and conduct of the study (applies to both Wellspect HealthCare staff and staff at the study site)
10. Previous enrolment or allocation of treatment in the present study.
11. Simultaneous participation in another clinical study that may interfere with the present study.
12. Severe non-compliance to protocol as judged by the investigator and/or Wellspect HealthCare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with bacteriuria <10^3 CFU/ml | 7 days
  Bacteriuria will be followed by daily urinary cultures, 3 hours after morning irrigation. The proportion of patients with at least one sample <10^3 CFU/ml within the 7 day treatment period will be evaluated.

SECONDARY OUTCOMES:
Time (number of days) to reduction of bacteriuria (<10^3 CFU/ml) | 7 days
  Bacteriuria will be followed by daily urinary cultures, 3 hours after morning irrigation. The number of days until reduction of bacteriuria (<10^3 CFU/ml) will be evaluated. Maximum treatment period is 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Rutberg, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (4):
- Sweden (4):
  - Spinal Cord Injury Unit, Sahlgrenska University Hospital, Gothenburg
  - Spinal Cord Injury Unit, Skåne University Hospital, Höör
  - Spinal Cord Injury Unit, Linköping University Hospital, Linköping
  - Neurocentrum, Neurorehab, Norrlands Universitetssjukhus, Umeå